CLINICAL TRIAL: NCT06773858
Title: Genetic Studies of Prostate Cancer Aggressiveness and Prognosis
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Fredrik Wiklund, Associate Professor, Karolinska Institutet
Other Study IDs: 2023-02626
Record Dates: First submitted 2025-01-02; First posted 2025-01-14 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Prostate Cancer (Adenocarcinoma); Prostate Cancer After a Radical Treatment
MeSH Terms: conditions — Prostatic Neoplasms; Adenocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- STHM3: A cohort comprising 2,295 men diagnosed with prostate cancer from the STHM3 trial population will be analyzed. Clinically significant disease is classified as cases with a Gleason grade ≥7, while aggressive disease is defined as stage T4 or cases with Gleason grade ≥8 in combination with stage T3. Indolent disease is characterized as cases with Gleason grade ≤6.

SUMMARY:
Prostate cancer is the most common form of cancer and the leading cause of cancer-related deaths among men in Sweden. In 2021, over 10,000 men were diagnosed with prostate cancer, and 2,077 died from the disease. Patients diagnosed with early-stage prostate cancer often undergo treatment aimed at curing the disease. However, since the side effects of active treatment are significant, it is crucial to identify new markers for aggressive forms of prostate cancer to better determine who would benefit most from curative treatment.

The investigators plan to conduct large-scale genetic studies using blood samples from men with prostate cancer. Specifically, the investigators will search for genetic markers associated with the development of more aggressive prostate cancer forms and markers for clinical progression. The clinical relevance of the identified genetic markers will be tested in a large population-based clinical prostate cancer study (the Stockholm-3 study).

The overall goal of this research is to discover new genetic markers for prostate cancer that may lead to more personalized and precise prostate cancer diagnostics.

DETAILED DESCRIPTION:
The investigators have the following specific aims:

Aim 1. To perform GWAS and create GRS for aggressive PCa A GWAS for aggressive PCa will be performed in international cohorts comprising 29,896 PCa patients (19,185 with non-aggressive disease and 10,711 with aggressive disease). Using summary statistics from this GWAS in a supervised machine learning framework, The investigators aim to create a GRS predictive of aggressive PCa.

Aim 2. To perform GWAS and create GRS for biochemical recurrence A GWAS for biochemical recurrence will be performed among patients who have undergone radical prostatectomy. Through international collaboration, 5,397 radical-operated patients will be available for assessment, among which biochemical recurrence occurred for 1,071 during follow-up. As in aim 1, supervised machine learning algorithms will be applied to the summary results from the GWAS to create a GRS for biochemical recurrence.

Aim 3. To perform a TWAS for aggressive disease and biochemical recurrence The investigators will perform a multi-tissue TWAS for aggressive disease and biochemical recurrence. Genetic prediction models will be trained using gene expression data measured in 22 tissues from over 3,900 individuals. Through these prediction models, gene expression levels will be imputed in the aggressive (aim 1) and biochemical recurrence (aim 2) study population and explored for association with disease aggressiveness and biochemical recurrence.

Aim 4. To assess the clinical translatability of GRS for aggressive disease and biochemical recurrence Using a large population-based Swedish clinical study of PCa detection, the clinical utility of GRS for aggressive disease and GRS for biochemical recurrence will be explored. In addition, a score based on rare pathogenic variants from 50 DNA repair genes will be assessed. The clinical utility of GRS will be established by comparing the added predictive performance of GRS above established predictive markers, PSA for detection, PSA, Gleason score, and TNM stage for a biochemical recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Living in Stockhol, Sweden
* Aged 50 to 69 years.

Exclusion Criteria:

* Previous diagnosis of prostate cancer

Ages: 50 Years to 69 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only men can develop prostate cancer.
Study Population: All men living in the Stockholm area, Sweden, aged 50 to 69 years.
Sampling Method: Non-Probability Sample
Enrollment: 2291 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Biochemical recurrence | From date of surgery date until the date of first documented recurrence or date of death from any cause, whichever came first, assessed up to 11 months
  According to American Urological Association guidelines, biochemical recurrence will be defined as a rise in PSA level of at least 0.2 ng/mL after surgery followed by a subsequent confirmatory PSA value of at least 0.2 ng/mL.

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska Institutet, Stockholm, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No
Only summary statistics from our study will be shared with other research groups to enable meta-analysis across groups.